CLINICAL TRIAL: NCT03778164
Title: Improving Prevention Systems to Reduce Disparities for High Priority Populations
Acronym: FastTrack
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Principal Investigator, Sarit Golub, Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH115835 (NIH)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: This study uses a cross sectional stepped wedge cluster randomized design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast Track Intervention (Experimental): This arm refers to the new Partner Services-Sexual Health intervention offered to contacts by the Partner Services program
  Interventions: Other: Fast Track Partner Services-Sexual Health Intervention
- Standard of Care (Active Comparator): This arm refers to the current standard practice for partners contacted by the Partner Services program
  Interventions: Other: Partner Services Standard of Care

INTERVENTIONS:
Other: Fast Track Partner Services-Sexual Health Intervention — The Partner Services-Sexual Health Intervention enhances the current standard of care by introducing four service innovations to the DOHMH Partner Services program: (1) enhanced field-based combination HIV and STI testing; (2) immediate field-based ARV/PrEP start; (3) navigation to a sexual health clinic for test results and treatment; and (4) enhanced linkage support to facilitate ongoing PrEP or HIV care.
  Arms: Fast Track Intervention
Other: Partner Services Standard of Care — Participants in neighborhoods that have not yet been assigned to the intervention condition in the stepped wedge trial will receive standard Partner Services components, including field-based HIV testing and referral to clinical sites for HIV prevention or treatment.
  Arms: Standard of Care

SUMMARY:
This project collaborates with the New York City Department of Health and Mental Hygiene (NYC DOHMH) to develop and test a field-based comprehensive sexual health intervention for HIV-exposed contacts notified by its Partner Services (i.e., HIV contact tracing) program. The goal of the study is to develop and test the impact of this new intervention on improving rates of HIV testing, linkage to HIV prevention/care, and PrEP uptake among highest risk contacts recently exposed to HIV. We will conduct a 6-month pilot project, followed by a cross-sectional stepped wedge cluster randomized trial in which 12 clusters of NYC neighborhoods are exposed to the intervention sequentially, with three clusters moving from control to intervention every 6 months (n = 1150). Primary outcomes are HIV testing, timely PrEP/ARV uptake, and linkage to PrEP/HIV care. Secondary outcomes are STD testing and receipt of STD treatment (if indicated).

ELIGIBILITY:
Inclusion Criteria:

* Contacts referred to the Partner Services program during the study time period

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1150 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Acceptance of HIV Testing | 1 month
  Whether or not contacts offered testing by the Partner Services program accept HIV testing
PrEP/ARV Initiation | 3 months
  Whether or not contacts start ARV medication in the field or at their referral visit
Linkage to PrEP/HIV Care | 6 months
  Whether or not contacts attend their navigation visit to receive ongoing PrEP or HIV services

SECONDARY OUTCOMES:
STI testing | 3 months
  Whether or not contacts accept STI testing in the field or at their referral visit

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter College of CUNY, New York, New York, United States